CLINICAL TRIAL: NCT05842590
Title: Clinical Evaluation of Direct Composite Veneer Restorations Performed in Permanent Incisors Affected by Molar-Incisor Hypomineralization
Brief Title: Clinical Evaluation of Direct Composite Veneer Restorations
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Hacettepe University (Other)
Responsible Party: Principal Investigator, Beste Ozgur, Assistant professor, Hacettepe University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HUDHF-Veneer
Record Dates: First submitted 2023-04-10; First posted 2023-05-06 (Actual); Last update posted 2023-05-06 (Actual); Status verified 2023-05

CONDITIONS: Molar Incisor Hypomineralization
MeSH Terms: conditions — Molar Hypomineralization

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Direct Composite Veneer (Experimental): This is a single-arm study. Direct composite veneer restoration will be performed to all patients.
  Interventions: Other: Composite Veneer Restoration

INTERVENTIONS:
Other: Composite Veneer Restoration — This is a single-arm study. Direct composite veneer Restorations will be performed to all patients.

SUMMARY:
The objective of this research was to evaluate the clinical success of direct composite veneer restorations performed in permanent incisors affected by molar-incisor hypomineralization.

ELIGIBILITY:
Inclusion Criteria:

* Cooperative children diagnosed with MIH according to European Academy of Paediatric Dentistry (EAPD) criteria
* Maxillary anterior teeth with MIH-caused coloring and opacity areas
* Fully erupted anterior teeth

Exclusion Criteria:

* Patients and parents of patients who accept to participate.
* Patients who are not in cooperation with the procedure.

Ages: 8 Years to 14 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 100 (Estimated)
Dates: Start 2022-08-02 (Actual); Primary Completion 2024-08 (Estimated); Study Completion 2024-08 (Estimated)

PRIMARY OUTCOMES:
1.Change from baseline to 12 months regarding "Anatomic form" | baseline, 3-month, 6-month,12-month
  alpha: The general contour of the restorations follows the contour bravo: the general contour of the restoration does not follow the contour of the tooth charlie: The restoration has an overhang does
2.Change from baseline to 12 months regarding "Marginal adaptation" | baseline, 3-month, 6-month,12-month
  alpha: Explorer does not catch or has one-way catch when drawn across the restoration/tooth interface bravo: explorer falls into crevice drawn across the restoration/tooth interface charlie: Dentin or base is exposed along the margin
3.Change from baseline to 12 months regarding "Surface roughness" | baseline, 3-month, 6-month,12-month
  alpha: the surface of the restoration does not have any surface defects bravo: the surface of the restoration has minimal surface defects charlie: the surface of the restoration has severe surface defects
4.Change from baseline to 12 months regarding "Marginal staining" | baseline, 3-month, 6-month,12-month
  alpha: there is no discoloration between the restorations and tooth bravo: there is discoloration on less than half of the circumferential margin charlie: there is discoloration on more than half of the circumferential margin
5.Change from baseline to 12 months regarding "Retention" | baseline, 3-month, 6-month,12-month
  alpha: intact bravo: chipped/loss of material charlie: complete loss of crown
6.Change from baseline to 12 months regarding "Incisal wear" | baseline, 3-month, 6-month,12-month
  alpha: intact bravo: wear of occlusal surface without tooth surface exposure charlie: wear of occlusal surface with tooth surface exposure

CONTACTS AND LOCATIONS:
Locations (1):
- Hacettepe University, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided